CLINICAL TRIAL: NCT01093365
Title: Effect of Varenicline on Cognitive Function in Cigarette Smokers With Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Tony George, Clinical Director, Schizophrenia Program, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 067/2009
Record Dates: First submitted 2010-03-24; First posted 2010-03-25 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Schizophrenia; Schizoaffective Disorder; Varenicline; Champix; Chantix; Nicotine; Nicotinic receptor; Dopamine; Acetylcholine; Cigarette; Smoking; Tobacco; Executive function; Working memory; Verbal memory; Cognitive function; Neuropsychological function
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Smoking | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Schizophrenia (Experimental): To measure the effects of varenicline on cognition of smokers with schizophrenia.
  Interventions: Drug: Varenicline

INTERVENTIONS:
Drug: Varenicline — * 0.0 mg orally twice per day for three days (placebo)
  * 0.5 mg orally twice per day for three days
  * 1.0 mg orally twice per day for three days
  Other Names: Chantix; Champix

SUMMARY:
Smokers with schizophrenia have more difficulties quitting smoking than smokers without a mental disorder. Varenicline (Champix) is a new stop smoking medication with a unique mechanism of action. It is a nicotine-like drug which is not addictive and not associated with the health risks of tobacco smoking.

Varenicline (VAR) binds to sites in the brain called nicotine receptors that play an important role in nicotine dependence. People with schizophrenia have difficulties in concentrating and remembering. Scientists believe that people with schizophrenia use smoking to remedy their cognitive problems. We will test VAR to see if it improves cognitive problems in smokers with schizophrenia in comparison to non-mentally ill smokers to determine whether people with schizophrenia get direct benefit from this nicotine-like drug. It is hypothesized that VAR (in comparison to a placebo) will reduce aspects of cognitive impairment in smokers and nonsmokers with schizophrenia.

DETAILED DESCRIPTION:
Schizophrenia is characterized by deficits in neurocognitive function, including executive function, attention, and spatial and verbal memory. Central nicotinic acetylcholine receptors (nAChR) are dysregulated in schizophrenia. It has been shown that neurocognitive deficits in schizophrenia improve by administration of nicotine, nicotinic agonists or cigarette smoking. Hence, it is believed that cigarette smoking may remedy cognitive deficits in schizophrenia and in fact some persons with schizophrenia may be "self-medicating" with tobacco to counter such cognitive problems.

The prevalence rates of cigarette smoking in persons with schizophrenia are higher than in the general population (58-88% vs. 25% respectively). This population also has a nicotine dependence rate of around 80 % and a high relapse rate after smoking cessation. Additionally the leading cause of medical problems and death in people with schizophrenia is tobacco addiction. Research that addresses the problem of smoking in schizophrenia is of great importance.

Varenicline (VAR), an α4β2 nAChR partial agonist, approved for smoking cessation, mimics the effect of nicotine by stimulating nAChRs, and releasing sufficient dopamine in order to reduce craving and withdrawal effects.

This study will follow four groups of subjects (N=40) that will receive neuropsychological and psychiatric testing in three consecutive sessions (smoking satiation, abstinence and reinstatement) separated by at least one week over 3 weeks. The groups are:

1. cigarette smokers with schizophrenia (N=10),
2. non-smokers with schizophrenia (N=10),
3. healthy cigarette smoking controls (N=10),
4. non-smoking controls (N=10).

All groups will be age- and sex- matched. Pre-treatment with varenicline (VAR) or placebo will start on Day 1 of each test session will be as follows: 1) 0.0 mg/day 2) 0.5 mg twice daily 3) or 1 mg twice daily for 3 days. Testing days will be separated by at least 1 week apart to rule out medication carry-over effects.

If nicotinic acetylcholine receptors can be stimulated resulting in more dopamine release and improved neurocognitive function without inducing deleterious health effects it may be of benefit to persons with schizophrenia who smoke tobacco.

ELIGIBILITY:
Inclusion Criteria:

I) For all subjects

* Age 18-55
* Estimated IQ ≥80 using the Shipley scale
* Capable of giving informed consent
* Not taking any form of nicotine replacement therapy

II) Additional inclusion criteria for smokers:

1. Non-treatment seeking cigarette smokers:

   * A score of 5 or higher on the Fagerstrom Test for Nicotine Dependence (FTND)
   * Self reported smoking of at least 10 cigarettes per day as measured by the Weekly Smoking Inventory (NOTE: Cigarette smoking is verified by a Smokerlyzer® test, with a cut off of 10 ppm and plasma cotinine levels ≥150 ng/ml)
2. Cigarette smokers with Schizophrenia:

   * Diagnosis of schizophrenia/schizoaffective disorder (confirmed by the SCID for DSM-IV)
   * Stable remission from positive symptoms of psychosis as judged by a score of <70 on the The Positive and Negative Syndrome Scale (PANSS) for schizophrenia and a psychiatric evaluation
   * Receiving a stable dose of antipsychotic medication(s)for the past month

III) Additional inclusion criteria for healthy smokers and non-smokers:

* No diagnosis for any Axis I psychiatric disorder (Except past history of major depression)

Exclusion Criteria:

For all subjects

* Substance abuse other than cigarette smoking.
* History of alcohol/drug abuse in the 3 months before study enrollment
* Hypersensitivity to varenicline (Champix)
* Use of opioids (meperidine, oxycodone, methadone, etc).
* A history of renal insufficiency
* Gastrointestinal problems including irritable bowel syndrome
* Exposure to chemotherapy
* A history of dementia and other neurological illness like epilepsy or medical condition known to significantly influence neurocognitive function
* Inability to learn the neuropsychological tasks during the training session
* Failure to demonstrate a deficit of at least 0.5 standard deviations below average levels of non-psychiatric control performance the on the Visuospatial Working Memory (VSWM) task
* Pregnancy
* Nursing women

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2010-03; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Computerized testing of neuropsychological functioning | Three times per week for three consecutive weeks
  * Trail Making Test, Part A
  * Trail Making Test, Part B
  * Visuospatial Working Memory (VSWM) and Digit Span of WAIS
  * Hopkins Verbal Learning Test - Revised (HVLT-V)
  * Continuous Performance Task (CPT)
Tiffany Urge to Smoke Scale | Three times per week for three consecutive weeks
Minnesota Withdrawal Scale | Three times over a two day period for three consecutive weeks

SECONDARY OUTCOMES:
Pre-pulse inhibition | 3 times per week for 3 weeks
  Measurement of startle reactivity to tones by EMG and the inhibition of the EMG response by exposure to a "pre-pulse".
Smoking topography | 3 times a week for 3 weeks
  Topographic assessment of smoking behavior (e.g., number of puffs per cigarette, puff volume, amount of time between puffs)

CONTACTS AND LOCATIONS:
Overall Officials: Tony P George, MD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health (33 Russell street), Toronto, Ontario, Canada

REFERENCES:
- [Derived] Johnstone S, Sorkhou M, Rabin RA, George TP. Dose-dependent effects of Varenicline on tobacco craving and withdrawal in tobacco smokers with and without schizophrenia. Drug Alcohol Depend. 2022 May 1;234:109412. doi: 10.1016/j.drugalcdep.2022.109412. Epub 2022 Mar 28. PMID 35395548
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching hospital. It is fully affiliated with the University of Toronto, and is a PAHO/WHO Collaborating Centre — http://www.camh.net/research